CLINICAL TRIAL: NCT01819961
Title: Randomized Clinical Trial of Omega-3 Fatty Acid-supplemented Parenteral Nutrition Versus Standard Parenteral Nutrition in Patients Undergoing Major Laparoscopic Abdominal Surgery
Brief Title: Parenteral Fish Oil in Major Laparoscopic Abdominal Surgery
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Wei Zhou (Other)
Responsible Party: Sponsor-Investigator, Wei Zhou, Attending, Sir Run Run Shaw Hospital
Organization: Sir Run Run Shaw Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Fo-Lap
Record Dates: First submitted 2013-03-20; First posted 2013-03-28 (Estimated); Last update posted 2013-03-28 (Estimated); Status verified 2013-03

CONDITIONS: Gastric Tumor; Pancreatic Tumor; Liver Tumor
MeSH Terms: conditions — Stomach Neoplasms; Pancreatic Neoplasms; Carcinoma, Hepatocellular | interventions — Fish Oils; fish oil triglycerides

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- MCT/LCT (Experimental): Structural Fat Emulsion Injection 250ml per day, for 7 days
  Interventions: Drug: MCT/LCT
- MCT/LCT and fish oil (Experimental): Structural Fat Emulsion Injection 250ml and fish oil 100ml for 7 days.
  Interventions: Drug: MCT/LCT and fish oil

INTERVENTIONS:
Drug: MCT/LCT and fish oil
  Other Names: Structural Fat Emulsion Injection (Fresenius-Kabi, Germany) and fish oil (Omegaven,Fresenius-Kabi, Germany)
  Arms: MCT/LCT and fish oil
Drug: MCT/LCT
  Other Names: Structural Fat Emulsion Injection (Fresenius-Kabi, Germany)
  Arms: MCT/LCT

SUMMARY:
The aim of this study is to assess the effect of postoperative parenteral fish oil on clinical outcome and immune function after major laparoscopic abdominal surgery.

DETAILED DESCRIPTION:
Postoperative patients are randomized by a sealed envelope to receive either a 50:50 (vol/vol) mixture of an oil rich in medium-chain fatty acids and soybean oil (termed MCT/LCT) or a mixture of MCT/LCT and fish oil Omegaven for 7 days. Full blood count, biochemistry and coagulation are routinely assessed. Fresh blood samples are centrifuged into plasma, red blood cells and lymphocytes then stored at -80°C pending analysis.

The primary endpoint was numbers of infective complications.Secondary endpoints were other clinical outcomes, length of hospital stay, and in-hospital mortality, along with plasma immunological markers.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing an elective major laparoscopic abdominal surgery and required at least 5 days of parenteral nutrition

Exclusion Criteria:

* Metabolic disease
* Chronic kidney or liver failure
* Shock
* Contraindications for lipid administration
* PN during the 15 days before hospitalisation

Ages: 15 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2013-04; Primary Completion 2013-10 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
infective complications | within the first 30 days after surgery

SECONDARY OUTCOMES:
length of hospital stay | average of 2 weeks
plasma immunological markers | from 1 day before surgery to 7 days after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Yiping Mou, MD, Study Director — Sir Run Run Shaw Hospital
Locations (1):
- Sir Run Run Shaw Hosptial, Hangzhou, Zhejiang, China